CLINICAL TRIAL: NCT01149551
Title: CSP #572 - Genetics of Functional Disability in Schizophrenia and Bipolar Illness
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 572
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; Bipolar disorder; Genetic research
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The purpose of this study is to detect genetic associations for the development of schizophrenia (SZ) and bipolar illness (BP) by comparing Veterans with these diseases to "psychiatrically healthy" Veterans from Veterans Health Administration medical centers. In addition, the genetic basis for functional capacity and disability in Veterans affected with SZ and BP will be assessed, as will genetic predictors of suicidality and tardive dyskinesia. Finally, we will also establish a repository which allows for future genomic studies related to SZ, BP, and related disorders or sequelae.

DETAILED DESCRIPTION:
We propose to identify the genetic basis of Veterans developing either of two major psychiatric (or "mental health") diseases: schizophrenia and bipolar disorder. The study will also examine the genetic basis of disability in everyday functions (such as employment, independent living, and self care) among the same patients. By "genetic basis," we mean how a person's genes might be a risk for developing these illnesses or being affected by them. We will compare information gathered from Veterans with these illnesses to "psychiatrically healthy" Veterans. Participants will be recruited from multiple Veterans Health Administration medical centers; the analysis of blood samples will be done in designated and approved laboratories.

Both schizophrenia and bipolar disorder are chronic psychiatric diseases associated with considerable lifelong disability; in particular, these illnesses are common in Veterans served by the Veterans Health Administration. Both of these conditions are also known to be caused in part by genes or so-called heredity; studies of the entire set of human genes (referred to as the genome) can be a tool to identify specific reasons why certain people develop certain conditions. In addition, patients with schizophrenia or bipolar disorder often have difficulty functioning in the real-world-including problems in attention and memory, or the ability to perform tasks of everyday living or have normal emotional experiences-and these "functional impairments" may also be inherited genetically. The current study is designed to help identify who is at higher risk for these diseases and related problems, so that better methods to diagnose and treat the conditions can be developed in the future.

Among other aspects of schizophrenia and bipolar disorder, suicide stands out as a very important issue to Veterans, their families, and the Veterans Health Administration. Suicide attempts and completed suicides are more common in Veterans with schizophrenia and bipolar illness (compared to Veterans without these illnesses), and this tendency may be inherited as well. Part of this study will involve determining whether specific genes might be associated with suicidal behavior. Similarly, the study will look at the genetic basis of side effects related to taking medications for these diseases.

For this research, participants will be recruited from VA sites that have extensive experience in conducting projects involving psychiatric disorders. We will collect information about the genes of these Veterans from a blood sample, and we will ask questions about health and related factors. We will also establish a repository which allows for future genomic studies related to SZ, BP, and related disorders or sequelae. The total study duration is indefinite in the setting of creating a SZ and BP repository, although the required time period for addressing the primary aims is 3.5 years. Data for a comparison ("reference") group of Veterans with medical, but not psychiatric, illnesses, will be obtained from a research initiative entitled the "VA Million Veteran Program" (VA-MVP).

Ultimately, this study attempts to advance the state-of-the-art regarding our understanding and treatment for two common mental health disorders affecting Veterans and will also serve as part of a major initiative to support "personalized" healthcare. It represents a major effort to link specific genes to illnesses, and eventually to treatments intended to relieve suffering.

ELIGIBILITY:
Inclusion Criteria:

Case participants:

* All participants must be 18 years of age or older
* SZ patients must meet lifetime (DSM-IV) criteria for schizophrenia, any subtype
* BP patients must have a confirmed bipolar type I diagnosis, which requires a history of a mixed or manic episode at some prior point, regardless of subsequent affective episodes
* all patients must have medical records available in the VA CPRS
* all patients must be competent to provide informed consent for the research

Control participants:

* Enrollment in the VA Million Veteran Program

Exclusion Criteria:

Case participants:

* SZ and BP patients that have participated in a previous GWAS study or are currently participating in a clinical treatment study
* patients with physical, sensory, or intellectual limitations that preclude their assessment with performance-based measures
* patients with active illicit drug use that might hamper assessments. Potential participants who present under the apparent influence of alcohol or drugs will be rescheduled once and excluded if they are intoxicated at their next appointment; patients identified via electronic medical record review will be screened for evidence of active drug abuse and excluded

Control participants:

* a personal history identifiable in the VA EMR of a major psychiatric disorder related to psychosis or a first degree family member with either schizophrenia or bipolar disorder
* major neurologic illnesses, or systemic medical illnesses, that could interfere with central nervous system function
* current treatment with psychotropic medications aimed at psychosis, bipolar disorder, or major depression
* anyone participating in an ongoing randomized trial of therapy for SZ or BP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case participants: Enrolled Veterans with a confirmed diagnosis of SZ and BP.
  Control participants: Psychiatrically healthy Veterans enrolled in VA Million Veteran Program.
Sampling Method: Non-Probability Sample
Enrollment: 9356 (Actual)
Dates: Start 2011-02; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Phenotypic cognitive and functional outcomes associated with SZ and BP | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip D. Harvey, PhD, Study Chair — Miami VA Healthcare System, Miami, FL
Locations (25):
- United States (25):
  - VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Central Arkansas VHS Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Brockton Campus, Brockton, MA, Brockton, Massachusetts
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas
  - VA Puget Sound Health Care System American Lake Division, Tacoma, WA, Tacoma, Washington